CLINICAL TRIAL: NCT02453724
Title: Lung Ultrasound Safety in Humans
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Vicki Noble, MD, Director, Division of Emergency Ultrasound, Massachusetts General Hospital
Other Study IDs: 2013P002671
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Pulmonary Hemorrhage
Keywords: Ultrasonography; Lung; Hemorrhage; Point of care ultrasound
MeSH Terms: conditions — Hemorrhage | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Observation for safety — The investigators will perform the routine lung exam used in emergency department evaluations for shortness of breath in patients scheduled for computed tomography. The investigators will observe if there are any parenchymal changes noted on the chest tomography scan.

SUMMARY:
The purpose of this study is to investigate if diagnostic ultrasound as it is routinely performed in humans causes lung hemorrhage significant enough to appear on thoracic CT. The investigators' hypothesis is that diagnostic lung ultrasound will not cause lung hemorrhage in humans. Damage to the lung in animal models has been shown to be mechanical rather than thermal in nature and evidence suggests that this injury is likely not from inertial cavitation but from alveolar resonance. Models of the alveolar resonance theory predict that hemorrhage should not happen in adult human lungs if the ultrasound frequency is higher than 1.69 MHz and mechanical index (MI) is less than 1.9 which is maintained with standard scanning protocol for thoracic ultrasound. A previous human study showed no gross macroscopic lung hemorrhage in patients undergoing transesophageal echocardiography with pressures of 2.4 MPa and MI 1.3 with exposure durations ranging 7-68 minutes.

The investigators propose to perform a routine lung ultrasound exam on patients who are scheduled to undergo chest computed tomography evaluation for pulmonary embolus as part of their routine care. The ultrasound will be performed immediately prior to CT imaging and markers will be placed on the patients chest to ensure the correct lung tissue is being evaluated. There will be two sham markers so the radiologist will be blinded to which tissue had ultrasound applied and which did not. The CT scan will then be evaluated per routine and also to see if there are signs of microscopic or macroscopic hemorrhage under the skin markers.

DETAILED DESCRIPTION:
This is a prospective, observational cohort study of emergency department patients designed to assess for radiographic changes suggestive of lung hemorrhage after thoracic ultrasound.

The investigators will only approach patients scheduled for CT scan as part of their routine care in the emergency department for enrollment. Only patients > 18 years old. Patients who are not english speaking will only be consented if there is a medical interpreter immediately available who can be approached for informed consent.

Patients who have given informed consent will have a lung ultrasound performed by a study physician immediately prior to CT scan - after the patient has been transported to the ED radiology area but before the CT scan is performed. The lung ultrasound will be performed using a low frequency probe (2-5 MHz). Of the four standard positions used in lung ultrasonography (Zone 1, 4, 5, 8; see Image 1 below), study ultrasonography will be performed on only two.

The two positions selected for use will be chosen immediately prior to ultrasound performance by the performing physician using a simple binary random number generator for each lung. This will ensure that one zone is subjected to ultrasound on each lung. A small radio-opaque button will be placed overlying all four zones (i.e., those exposed and those not exposed) in the standard position of the ultrasound footprint (ie where the ultrasound was or would have been performed) and then the patient will undergo the CT scan according to standard radiology department protocols.

The CT scan will then be reviewed for signs of alveolar hemorrhage in the lung tissue immediately adjacent to the radio-opaque button. Radiologists will be blinded as to which buttons abut zones exposed to ultrasound or not exposed. Any findings will be immediately reported to the patient's care team and the patient and standard protocols for treatment and observation will be followed.

The investigators have calculated the need to enroll 200 patients to observe a 7% range above and below previously published numbers of incidental findings on chest CT scan.

ELIGIBILITY:
Inclusion Criteria:

* All patients greater than 18 years of age scheduled to receive chest tomography scans for pulmonary embolus.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All emergency department patients greater than 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Micro or macroscopic lung parenchymal hemorrhage | At enrollment
  The investigators will perform the ultrasound just prior to chest computed tomography enrollment so that there is minimal time delay between the ultrasound performance and assessment of the lung parenchyma.

CONTACTS AND LOCATIONS:
Overall Officials: Vicki E Noble, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] O'Brien WD Jr, Yang Y, Simpson DG, Frizzell LA, Miller RJ, Blue JP Jr, Zachary JF. Threshold estimation of ultrasound-induced lung hemorrhage in adult rabbits and comparison of thresholds in mice, rats, rabbits and pigs. Ultrasound Med Biol. 2006 Nov;32(11):1793-804. doi: 10.1016/j.ultrasmedbio.2006.03.011. PMID 17112965
- [Background] Miller DL. Induction of pulmonary hemorrhage in rats during diagnostic ultrasound. Ultrasound Med Biol. 2012 Aug;38(8):1476-82. doi: 10.1016/j.ultrasmedbio.2012.04.004. Epub 2012 Jun 12. PMID 22698500
- [Background] Jabaraj DJ, Jaafar MS. Theoretical calculation of resonant frequencies of the human alveolar wall and its implications in ultrasound-induced lung hemorrhage. Int J Bioscience Biochem Bioinformatics. 2013;3(1):5-9
- [Background] Meltzer RS, Adsumelli R, Risher WH, Hicks GL Jr, Stern DH, Shah PM, Wojtczak JA, Lustik SJ, Gayeski TE, Shapiro JR, Carstensen EL. Lack of lung hemorrhage in humans after intraoperative transesophageal echocardiography with ultrasound exposure conditions similar to those causing lung hemorrhage in laboratory animals. J Am Soc Echocardiogr. 1998 Jan;11(1):57-60. doi: 10.1016/s0894-7317(98)70120-8. PMID 9487470
- [Background] Bruzzi JF, Remy-Jardin M, Delhaye D, Teisseire A, Khalil C, Remy J. Multi-detector row CT of hemoptysis. Radiographics. 2006 Jan-Feb;26(1):3-22. doi: 10.1148/rg.261045726. PMID 16418239
- [Result] Child SZ, Hartman CL, Schery LA, Carstensen EL. Lung damage from exposure to pulsed ultrasound. Ultrasound Med Biol. 1990;16(8):817-25. doi: 10.1016/0301-5629(90)90046-f. PMID 2095012